CLINICAL TRIAL: NCT04153409
Title: A Proof of Concept Study of the Efficacy and Safety of Oral LAT8881 in Acute Migraine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lateral Pharma Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LAT-MIG-001
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Results first posted 2021-03-30 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Acute Migraine

STUDY DESIGN:
Intervention Model Description: Randomised assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Active (Experimental): Subjects will be given two 30 mg capsules of the investigational medicinal product (LAT8881), and instructed to take both capsules within the first hour of the onset of a migraine of moderate to severe intensity.
  Interventions: Drug: LAT8881
- Placebo (Placebo Comparator): Subjects will be given two capsules of placebo, and instructed to take both capsules within the first hour of the onset of a migraine of moderate to severe intensity.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LAT8881 — Two 30 mg capsules of LAT8881
  Arms: Active
Drug: Placebo — Two capsules of placebo
  Arms: Placebo

SUMMARY:
This is a randomised, placebo controlled, double blind, crossover proof of concept study to investigate the efficacy and safety of oral LAT8881 in acute migraine, with or without aura.

DETAILED DESCRIPTION:
Subjects enrolled in the study will be randomised to receive investigational medicinal product (LAT8881 60 mg or placebo), to be taken at the onset (within one hour from the onset of pain) of a migraine headache of moderate to severe intensity [Numeric rating scale greater than 4]. Rescue medication should not be taken until at least 2 hours post dose. Subjects will be given a single dose of either active or placebo, to treat one migraine headache.

After treatment of one migraine headache (or a maximum 28 days) the subject will return to the clinic for re-evaluation and crossover to the second treatment. After treatment of one migraine headache in the second treatment period or a maximum of 28 days from commencement of the second treatment period, the subject will return to the clinic for re-evaluation. An End of study visit (telephone) will occur 7 days after the end of the second treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 18 to 75 years at the time of consent
2. Diagnosis of episodic migraine headache at least 12 months ago with or without aura as defined in International Classification of Headache-3
3. Onset of migraine headache before age 50
4. Medical history of 2 - 8 migraine headache attacks per month for the previous 12 months; ≥ 75% of attacks progress to moderate or severe pain within 2 hours (ie, rapidly-escalating)
5. Minimum 48 hours on average between migraine headache attacks
6. Acute headache medication on ≤ 14 days/month in the 3 months prior to screening
7. Willing and able to comply with all study procedures including completion of a headache diary and a migraine diary on the day of a migraine headache

Exclusion Criteria:

1. Unable to distinguish migraine from other primary headache conditions
2. Average of 15 or more headache (migraine or nonmigraine) days per month or history of more than 25% of headaches occurring at time of wakening (wake up headaches)
3. History of aura lasting more than 60 minutes
4. History of vomiting within 2 hours of onset of a migraine headache in more than 25% of migraine headaches
5. Medication overuse headache, defined as:

   1. use of opioids, triptans or ergot alkaloids or any combination of these medications for treatment of headaches 10 or more days per month during the 90 days prior to screening OR
   2. Non-steroidal anti-inflammatory drugs (NSAIDs) or simple analgesics for treatment of headaches on more than 14 days per month during the 90 days prior to screening
6. Recent (3 years) history of frequent or chronic hemiplegic/ basilar migraine, tension headache, retinal migraine, ophthalmoplegic migraine as per ICHD classification, or treatment resistant atypical migraine
7. Hospital admission for status intractable migraine or medication overuse headache within 6 months of screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-04-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - Paratus Clinical Research, Central Coast, Kanwal, New South Wales
  - Paratus Clinical Research, Blacktown, Sydney, New South Wales
  - Emeritus Research, Camberwell, Victoria

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- LAT8881, Then Placebo: Subjects took LAT8881 60 mg (2 capsules) at the onset of a migraine of moderate to severe intensity. After treatment of one migraine (or a maximum of 28 days), subjects took 2 placebo capsules at the onset of a migraine of moderate to severe intensity.
- Placebo, Then LAT8881: Subjects took 2 placebo capsules at the onset of a migraine of moderate to severe intensity. After treatment of one migraine (or a maximum of 28 days), subjects took LAT8881 60 mg (2 capsules) at the onset of a migraine of moderate to severe intensity.
Period: Overall Study
Arm/Group | LAT8881, Then Placebo | Placebo, Then LAT8881
Started | 10 | 11
Completed | 8 | 9
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LAT8881, Then Placebo | Placebo, Then LAT8881 | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (9.61) | 41.2 (13.64) | 40.0 (11.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 11 | 21
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Australia | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change in Migraine Headache Pain Score From Time of Dosing (0 Minutes)
Description: Change in migraine headache pain score, using an 11-point numeric rating scale (NRS), (0 = none, 10 = worst imaginable), Pain is recorded in a subject diary and should reflect the subject's pain at the time of recording. A reduction in NRS score indicates a reduction in pain intensity.
Time Frame: 0 minutes, 30 minutes, 60 minutes, 90 minutes, 2 hours, 4 hours, 8 hours and 24 hours post dose
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active | Placebo
Number analyzed (Participants) | 16 | 17
score on a scale
  Change from baseline at 0.5 hours | 0 (1.10) | 0.2 (1.33)
  Change from baseline at 1 hour | -0.8 (1.83) | -0.2 (1.68)
  Change from baseline at 1.5 hours | -0.9 (2.36) | -0.5 (1.84)
  Change from baseline at 2 hours | -1.8 (3.12) | -0.8 (2.63)
  Change from baseline at 4 hours | -2.7 (2.96) | -2.2 (3.56)
  Change from baseline at 8 hours | -4.6 (2.31) | -3.7 (3.39)
  Change from baseline at 24 hours | -5.8 (1.87) | -5.6 (2.8)
Statistical Analysis 1: Comparison: Active vs Placebo; Change from baseline at 0.5 hours; Test type: Superiority — No formal sample size estimation was undertaken due to the exploratory nature of the study. Statistical comparisons of the 7 mean changes from baseline to different time-points (0-24 hours) were undertaken in one mixed effects model of analysis taking into account the cross-over nature of the study and the multiple time points within each period to explore a possible treatment effect in this small proof of concept study. Change from baseline at 0.5 hours is presented in this section; p = 0.9733, Mixed Models Analysis — No adjustment for multiple comparisons has been made due to the exploratory nature of the study; Mean Difference (Net) = -0.02, 95% CI 2-sided [-1.23 to 1.19] — Difference is Active-Placebo
Statistical Analysis 2: Comparison: Active vs Placebo; Change from baseline at 1 hour. The change from baseline at 1 hour was extracted from the mixed model analysis including all time points; Test type: Superiority; p = 0.4942, Mixed Models Analysis — No adjustment for multiple comparisons has been made due to the exploratory nature of the study; Mean Difference (Net) = -0.42, 95% CI 2-sided [-1.64 to 0.79] — Difference is Active-Placebo
Statistical Analysis 3: Comparison: Active vs Placebo; Change from baseline at 1.5 hours. The change from baseline at 1.5 hours was extracted from the mixed model analysis including all time points; Test type: Superiority; p = 0.6866, Mixed Models Analysis — No adjustment for multiple comparisons has been made due to the exploratory nature of the study; Mean Difference (Net) = -0.25, 95% CI 2-sided [-1.46 to 0.97] — Difference is Active-Placebo
Statistical Analysis 4: Comparison: Active vs Placebo; Change from baseline at 2 hours. The change from baseline at 2 hours was extracted from the mixed model analysis including all time points; Test type: Superiority; p = 0.1488, Mixed Models Analysis — No adjustment for multiple comparisons has been made due to the exploratory nature of the study; Mean Difference (Net) = -0.89, 95% CI 2-sided [-2.11 to 0.32] — Difference is Active-Placebo
Statistical Analysis 5: Comparison: Active vs Placebo; Change from baseline at 4 hours. The change from baseline at 4 hours was extracted from the mixed model analysis including all time points; Test type: Superiority; p = 0.5644, Mixed Models Analysis — No adjustment for multiple comparisons has been made due to the exploratory nature of the study; Mean Difference (Net) = -0.36, 95% CI 2-sided [-1.57 to 0.86] — Difference is Active-Placebo
Statistical Analysis 6: Comparison: Active vs Placebo; Change from baseline at 8 hours, The change from baseline at 8 hours was extracted from the mixed model analysis including all time points; Test type: Superiority; p = 0.2561, Mixed Models Analysis — No adjustment for multiple comparisons has been made due to the exploratory nature of the study; Mean Difference (Net) = -0.70, 95% CI 2-sided [-1.91 to 0.51] — Difference is Active-Placebo
Statistical Analysis 7: Comparison: Active vs Placebo; Change from baseline at 24 hours. The change from baseline at 24 hours was extracted from the mixed model analysis including all time points; Test type: Superiority; p = 0.9875, Mixed Models Analysis — No adjustment for multiple comparisons has been made due to the exploratory nature of the study; Mean Difference (Net) = -0.01, 95% CI 2-sided [-1.22 to 1.20] — Difference is Active-Placebo

2. Secondary Outcome: Change in Migraine-associated Symptoms of Nausea, Photophobia and Phonophobia From Time of Dosing (0 Minutes)
Description: Symptoms are assessed on an 11- point Likert scale (0 = no symptoms, 10 = severe symptoms). A larger negative number represents a greater reduction in symptom intensity
Time Frame: 0 minutes, 30 minutes, 60 minutes, 90 minutes, 2 hours, 4 hours, 8 hours and 24 hours post dose
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active | Placebo
Number analyzed (Participants) | 16 | 17
score on a scale
  Change in nausea at 0.5 hours | -0.3 (2.24) | -0.1 (1.05)
  Change in nausea at 1 hour | -0.9 (2.87) | -0.6 (1.28)
  Change in nausea at 1.5 hours | -1.0 (3.93) | -1.0 (1.70)
  Change in nausea at 2 hours | -1.6 (4.02) | -1.0 (2.00)
  Change in nausea at 4 hours | -2.1 (4.30) | -2.1 (2.41)
  Change in nausea at 8 hours | -4.3 (3.32) | -2.8 (3.60)
  Change in nausea at 24 hours | -4.9 (3.04) | -3.6 (2.89)
  Change in photophobia at 0.5 hours | -0.2 (0.75) | 0.2 (1.07)
  Change in photophobia at 1 hour | -0.9 (1.91) | 0.0 (1.46)
  Change in photophobia at 1.5 hours | -0.8 (2.08) | -0.8 (2.59)
  Change in photophobia at 2 hours | -1.3 (2.52) | -0.9 (2.93)
  Change in photophobia at 4 hours | -2.1 (2.70) | -2.4 (3.68)
  Change in photophobia at 8 hours | -3.8 (2.52) | -3.6 (3.54)
  Change in photophobia at 24 hours | -4.6 (2.39) | -4.4 (3.12)
  Change in phonophobia at 0.5 hours | 0.1 (0.89) | -0.2 (1.68)
  Change in phonophobia at 1 hour | -0.6 (2.09) | -0.4 (1.73)
  Change in phonophobia at 1.5 hours | -0.5 (2.19) | -0.8 (1.95)
  Change in phonophobia at 2 hours | -0.2 (2.61) | -0.7 (2.31)
  Change in phonophobia at 4 hours | -0.6 (2.53) | -1.8 (3.05)
  Change in phonophobia at 8 hours | -1.8 (2.48) | -2.3 (2.91)
  Change in phonophobia at 24 hours | -2.3 (2.35) | -2.6 (2.89)

3. Secondary Outcome: Change in Each Subject's Most Troublesome Symptom From Time of Dosing (0 Minutes)
Description: as for outcome 2
Time Frame: 0 minutes, 30 minutes, 60 minutes, 90 minutes, 2 hours, 4 hours, 8 hours and 24 hours post dose
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active | Placebo
Number analyzed (Participants) | 16 | 17
score on a scale
  Change from baseline at 0.5 hours | -0.5 (2.03) | -0.1 (1.60)
  Change from baseline at 1 hour | -1.1 (2.33) | -0.6 (2.06)
  Change from base at 1.5 hours | -1.2 (3.06) | -1.2 (2.86)
  Change from baseline at 2 hours | -1.5 (3.46) | -1.5 (3.16)
  Change from baseline at 4 hours | -2.6 (3.58) | -2.8 (3.68)
  Change from baseline at 8 hours | -3.9 (2.69) | -4.0 (3.26)
  Change from baseline at 24 hours | -5.2 (2.01) | -5.0 (2.78)

4. Secondary Outcome: The Percentage of Subjects Achieving "no Headache Pain"
Description: Defined as having no migraine headache pain
Time Frame: 30 minutes, 60 minutes, 90 minutes, 2 hours, 4 hours, 8 hours post-dose
Population: Per protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Active | Placebo
Number analyzed (Participants) | 16 | 17
Participants
  0.5 hours | 0 | 0
  1 hour | 0 | 0
  1.5 hours | 0 | 0
  2 hours | 2 | 0
  4 hours | 2 | 2
  8 hours | 6 | 6
  24 hours | 11 | 12

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the first dose until the end of study visit, approximately 64 days
Arm/Group | Active | Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 3/17 | 3/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=17) | Placebo (N=17)
Otitis externa (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Except for legal reasons, the investigator will not reveal the result of the study to a third party without a mutual agreement about the analysis and interpretation of the data with the sponsor.

DOCUMENTS (2):
  • Study Protocol (2019-07-25): https://cdn.clinicaltrials.gov/large-docs/09/NCT04153409/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-27): https://cdn.clinicaltrials.gov/large-docs/09/NCT04153409/SAP_001.pdf